CLINICAL TRIAL: NCT00528905
Title: A Multi-Center Randomized, Placebo-Controlled, Double-Blind, Parallel Group, Phase IIb Proof of Concept Study With 3 Oral Groups of AZD3480 During 12 Weeks Treatment of Cognitive Deficits in Patients With Schizophrenia
Brief Title: Proof of Concept Study of Cognitive Improvement in Patients With Schizophrenia
Acronym: HALO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D3690C00011
Record Dates: First submitted 2007-09-10; First posted 2007-09-12 (Estimated); Last update posted 2008-11-25 (Estimated); Status verified 2008-11

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Cognitive Deficits
MeSH Terms: conditions — Schizophrenia; Cognition Disorders | interventions — ispronicline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Placebo Comparator): Placebo
  Interventions: Drug: AZD3480
- 2 (Experimental): AZD3480 oral
  Interventions: Drug: AZD3480
- 3 (Experimental): AZD3480 oral dose
  Interventions: Drug: AZD3480

INTERVENTIONS:
Drug: AZD3480 — oral capsule

SUMMARY:
The purpose of this study is to demonstrate that AZD3480 improves cognition in patients with stable schizophrenia who are being treated with an atypical antipsychotic and who are active cigarette smokers, to assess the safety and tolerability of AZD3480 and to define the optimal dose(s) to be used in future trials.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia
* Outpatient at the time of screening and randomization
* Stable housing defined as having a place to live in the community (ie, not in a hospital or nursing home)
* Active cigarette smoking (10 or more cigarettes per day

Exclusion Criteria:

* Any significant psychiatric or neurological disease other than schizophrenia, or current diagnosis of major depressive disorder
* Known or suspected drug or alcohol abuse within the 6 months or urine toxicology test positive for illegal or non-prescribed substances
* Impaired vision and/or hearing making cognitive testing difficult

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 400 (Estimated)
Dates: Start 2007-08; Primary Completion 2008-10 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Domain scores for Attention/Vigilance, Working Memory, Verbal Learning, Speed of Processing and Verbal Fluency as measured on the IntegNeuro computerized test battery of cognitive function | Change from baseline to Week 12

SECONDARY OUTCOMES:
UCSD Performance Based Skills Assessment (UPSA2) and on the Social Functioning Scale (SFS) | Change from baseline to Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Larry Rodichok, MD, Study Director — AstraZeneca
Locations (80):
- United States (66):
  - Research Site, Little Rock, Arkansas
  - Research Site, Anaheim, California
  - Research Site, Cerritos, California
  - Research Site, Costa Mesa, California
  - Research Site, Escondido, California
  - Research Site, Garden Grove, California
  - Research Site, Long Beach, California
  - Research Site, Los Angeles, California
  - Research Site, Oceanside, California
  - Research Site, Pasadena, California
  - Research Site, Pico Rivera, California
  - Research Site, San Diego, California
  - Research Site, Santa Ana, California
  - Research Site, New Britain, Connecticut
  - Research Site, New Haven, Connecticut
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Boca Raton, Florida
  - Research Site, Coral Gables, Florida
  - Research Site, North Miami, Florida
  - Research Site, Orlando, Florida
  - Research Site, Tampa, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Augusta, Georgia
  - Research Site, Marietta, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Joliet, Illinois
  - Research Site, Schaumburg, Illinois
  - Research Site, Indianapolis, Indiana
  - Research Site, New Orleans, Louisiana
  - Research Site, Glen Burnie, Maryland
  - Research Site, Haverhill, Massachusetts
  - Research Site, Pittsfield, Massachusetts
  - Research Site, Minneapolis, Minnesota
  - Research Site, St Louis, Missouri
  - Research Site, Las Vegas, Nevada
  - Research Site, Nashua, New Hampshire
  - Research Site, Cherry Hill, New Jersey
  - Research Site, Clementon, New Jersey
  - Research Site, East Orange, New Jersey
  - Research Site, Newark, New Jersey
  - Research Site, Paramus, New Jersey
  - Research Site, Brooklyn, New York
  - Research Site, Cedarhurst, New York
  - Research Site, Elmsford, New York
  - Research Site, Glen Oaks, New York
  - Research Site, Jamaica, New York
  - Research Site, New York, New York
  - Research Site, Rochester, New York
  - Research Site, Staten Island, New York
  - Research Site, Cincinnati, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Kettering, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Allentown, Pennsylvania
  - Research Site, DuBois, Pennsylvania
  - Research Site, Norristown, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Charleston, South Carolina
  - Research Site, Memphis, Tennessee
  - Research Site, Austin, Texas
  - Research Site, DeSoto, Texas
  - Research Site, Houston, Texas
  - Research Site, Irving, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Richmond, Virginia
  - Research Site, Spokane, Washington
- Canada (14):
  - Research Site, Calgary, Alberta
  - Research Site, Red Deer, Alberta
  - Research Site, Penticton, British Columbia
  - Research Site, Victoria, British Columbia
  - Research Site, Winnipeg, Manitoba
  - Research Site, Halifax, Nova Scotia
  - Research Site, Sydney, Nova Scotia
  - Research Site, Burlington, Ontario
  - Research Site, Greater Sudbury, Ontario
  - Research Site, Mississauga, Ontario
  - Research Site, Orléans, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Windsor, Ontario
  - Research Site, Montreal, Quebec